CLINICAL TRIAL: NCT06324201
Title: The Long-term Safety and Effectiveness Evaluation of the QDOT MICRO™ System Use in Conjunction With VISITAG SURPOINT™Module for the Treatment of Symptomatic Drug Refractory Paroxysmal Atrial Fibrillation
Brief Title: The Long-term Safety and Effectiveness Evaluation of the QDOT MICRO System Use in Conjunction With VISITAG SURPOINT Module for the Treatment of Symptomatic Drug Refractory Paroxysmal Atrial Fibrillation.
Acronym: QDOT PAS
Status: Recruiting | Type: Observational
Sponsor: Heart Rhythm Clinical and Research Solutions, LLC (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: QDOT PAS
Record Dates: First submitted 2024-02-21; First posted 2024-03-21 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ablation Procedure — Ablation Procedure for paroxysmal atrial fibrillation

SUMMARY:
Observational, multi-center, non-randomized, post-market study. This is a nested sub-study of the REAL AF Registry. Consecutive symptomatic drug refractory paroxysmal atrial fibrillation (PAF) patients from the registry will be screened for enrollment, prospectively or retrospectively, to this sub-study per inclusion and exclusion criteria.

DETAILED DESCRIPTION:
Enrolled QDOT PAS subjects are defined as consented patients with symptomatic paroxysmal atrial fibrillation (PAF) enrolled in the REAL AF registry. These enrolled subjects will be treated with the commercially available QDOT MICRO™ system (QDOT MICRO™ catheter and nGEN™ generator) in conjunction with VISITAG SURPOINT™ Module. Subjects are required to complete scheduled assessments within 12 months of the index procedure, and additional two assessments at 24 and 36-months post procedure. Retrospective consecutive patients from the REAL AF registry, who were ablated with the QDOT MICRO™ system, may be enrolled into the sub-study if the patient meets eligibility criteria and provides consent for additional follow-up of 24 and 36-months

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic drug refractory paroxysmal (AF episode terminate spontaneously within 7 days) who, in the opinion of the investigator, are candidates for ablation for AF
2. 18 years of age or older
3. Able and willing to participate in baseline and follow up evaluations for the full length of the sub-study
4. Willing and able to provide informed consent for this sub-study

Exclusion Criteria:

1. Patients who have undergone catheter ablation for atrial fibrillation (PVI, roof line, posterior wall ablation...)
2. Enrolled in an investigational drug or device clinical trial, or any trial that dictates the treatment plan
3. Persistent or long-standing persistent AF
4. In the opinion of the investigator, any known contraindication to an ablation procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will consist of patients in the REAL AF registry who have symptomatic PAF and will have, or have undergone, ablation procedures using the QDOT MICRO™ System with VISITAG SURPOINT™ Module
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Safety of the QDOT Micro System use in conjunction with VISITAG SURPOINT Module | Day 0-7 post ablation
  Adverse events from post-procedure through 7-day post ablation visit.
Effectiveness of the QDOT Micro System use in conjunction with VISITAG SURPOINT Module at 12-months. | 12 months
  Freedom from atrial arrhythmia recurrence at 12 months post procedure.
Effectiveness of the QDOT Micro System use in conjunction with VISITAG SURPOINT Module at 24-months. | 24 months
  Freedom from atrial arrhythmia recurrence at 24 months post procedure.
Effectiveness of the QDOT Micro System use in conjunction with VISITAG SURPOINT Module at 36-months. | 36 months
  Freedom from atrial arrhythmia recurrence at 36 months post procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Sanchez, MD, Study Director — J & J Corporation
Locations (21):
- United States (21):
  - Arrhythmia Institute at Grandview, Birmingham, Alabama
  - Mobile Cardiology Associates, Mobile, Alabama
  - Community Memorial Health System, Ventura, California
  - Medical City - HCA, Aurora, Colorado
  - Naples Community Hospital, Naples, Florida
  - Sarasota Memorial Health, Sarasota, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - Norton Heart and Vascular Institute, Louisville, Kentucky
  - The Brigham and Womens Hospital, Boston, Massachusetts
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Trinity Health-Michigan Heart, Ypsilanti, Michigan
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pennsylvania (UPENN), Philadelphia, Pennsylvania
  - Allegheny Health, Pittsburgh, Pennsylvania
  - Centra Health, Inc.dba Stroobants Cardiovascular Center, Lynchburg, Virginia
  - Bon Secours Medical Group - Richmond Specialty Care, Richmond, Virginia
  - Valley Health System, Winchester, Virginia
  - Multicare Health Systems-Pulse Heart, Puyallup, Washington
  - Franciscan Heart and Vascular Associates, Tacoma, Washington
  - Mercy Health, Janesville, Wisconsin

IPD SHARING:
Plan to Share IPD: No